CLINICAL TRIAL: NCT00990132
Title: Randomised Controlled Trial of Home Mechanical Ventilation in Hypercapnic Chronic Obstructive Pulmonary Disease Patients Post Acute Hypercapnic Exacerbation
Brief Title: Home Mechanical Ventilation vs Home Oxygen Therapy in COPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Patrick Murphy (Other)
Collaborators: Guy's & St Thomas' Charity (Other); Respironics International (Industry); ResMed (Industry); ResMed Foundation (Other)
Responsible Party: Sponsor-Investigator, Patrick Murphy, PI, Guy's and St Thomas' NHS Foundation Trust
Organization: Guy's and St Thomas' NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ1 09/N070
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Respiratory failure; Non-invasive ventilation; Home mechanical ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long term oxygen therapy (Active Comparator): LTOT will be established as per current national guidelines
  Interventions: Device: Long term oxygen therapy
- Home mechanical ventilation (Experimental): Patients will be set up on LTOT as per national guidelines and nocturnal non-invasive ventilation in accordance with study protocol.
  Interventions: Device: Home mechanical ventilation

INTERVENTIONS:
Device: Home mechanical ventilation — Nocturnal non-invasive ventilation
  Other Names: Harmony 2; VPAP III STA
  Arms: Home mechanical ventilation
Device: Long term oxygen therapy — LTOT established as per national guidelines
  Arms: Long term oxygen therapy

SUMMARY:
This study is designed to investigate the effect of home mechanical ventilation (HMV) in patients with severe chronic obstructive pulmonary disease (COPD). The purpose of the trial is to test the hypothesis that HMV and longterm oxygen therapy (LTOT) increases admission free survival compared with LTOT alone. More specifically, compared with LTOT, HMV and LTOT reduces hospital re-admission in COPD patients who remain persistently hypercapnic following an acute exacerbation requiring non-invasive ventilation (NIV).

DETAILED DESCRIPTION:
Although HMV has been shown to improve physiological parameters as well as have clinical benefits in terms of dyspnoea and exercise capacity in severe COPD, the published randomised controlled trials have been less positive. The Steering Committee are committed to design a robust clinical trial that will answer this clinical question. Therefore, a multi-centre randomised controlled trial has been designed with recruitment and power calculations based on the applicants own data.

We will recruit from 8 UK university centres with expertise in HMV, 116 hypercapnic patients (58 in each arm) with persistent hypercapnia following an episode of acute hypercapnic respiratory failure. During the acute hypercapnic episode the patient would have be eligible for non-invasive ventilation with a pH <7.35 and a partial pressure of carbon dioxide (PaCO2) > 7.0kPa. They will be randomised, for a 12 months, to either

1. HMV and LTOT (Treatment Group)
2. LTOT alone (Control Group) This study would allow the investigators to answer a number of questions pertaining to clinical efficacy of HMV in COPD as well as the mechanism of action of HMV in COPD

   * Does HMV effect admission-free survival?
   * Does HMV reduce exacerbation frequency?
   * Does HMV impact on disease progression?
   * Does HMV improve health-related quality of life?
   * Does HMV improve exercise capacity?
   * Is there a dose-response between hours of ventilator compliance and daytime PaO2 and PaCO2?
   * Do patients increase hours of ventilator use during acute exacerbations?
   * Is ventilator compliance with HMV and LTOT acceptable?
   * Does HMV reduce healthcare utilisation? Follow-up assessments will be performed at 6 weeks, 3, 6 and 12 months. These data collected will include admission-free survival (primary outcome), hours of compliance with HMV, HRQL, gas exchange, lung function, body composition, exercise capacity, exacerbation frequency primary care consultations and compliance with LTOT, time to withdrawal of LTOT/night-time oxygen therapy based on daytime PaO2 and overnight SaO2 (secondary outcome measures). The relation of any changes to factors predicting severity of COPD will be studied. The cost effectiveness and cost-utility analysis of HMV will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD
* Acute hypercapnic exacerbation of COPD at least 2 weeks previously
* Tolerated non-invasive ventilation during acute hypercapnic exacerbation
* Chronic hypoxia requiring LTOT (PaO2 <7.3kPa or a PaO2 >7.3 and <8.0kPa and one of the following: secondary polycythaemia; nocturnal hypoxaemia SaO2 <90% for >30% of the time; peripheral oedema; or PHT)
* Chronic hypercapnia (PaCO2 >7kPa)
* ≥20 pack year smoking history
* FEV1/FVC <60%
* FEV1 at <50% predicted

Exclusion Criteria:

* Persistent hypercapnic respiratory failure with acidosis (defined as pH <7.30 after bronchodilators)
* Development of worsening hypercapnic respiratory failure with acidosis during initiation of LTOT therapy
* Failure to tolerate NIV during the acute illness preceding trial identification
* Post extubation or decannulation following AHRF requiring intubation
* Restrictive lung disease causing hypercapnia i.e. obesity hypoventilation and chest wall disease, however these patients will be included if the FEV1/FVC ratio is <60% and the FEV1 <50% if the predominant defect is considered to be obstructive by the center clinician.
* Clinical features of severe OSA
* BMI >35kg/m2
* Unstable coronary artery syndrome
* Cognitive impairment that would prevent informed consent into the trial
* Psychiatric disease necessitating anti-psychotic medication, ongoing treatment for drug or alcohol addiction, persons of no fixed abode post-discharge
* Patients undergoing renal replacement therapy
* Age <18 years
* Pregnant
* Inability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Days from trial intervention to either hospital admission or death | 1 year

SECONDARY OUTCOMES:
Spirometry - specifically FEV1 & FVC change from trial intervention to follow up. | 1 year
Changes Health related quality of life from pre-intervention to follow up - specifically outcomes of severe respiratory insufficiency questionnaire, chronic respiratory disease questionnaire & MRC dyspnoea score | 1 year
Change in arterial PaCO2 from pre-intervention to follow up | 1 year
Change in the incremental shuttle walk test from pre-intervention to follow up | 1 year
Frequency of acute exacerbations of COPD requiring addition of antibiotics and or steroids and or hospital admission | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Murphy, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Nicholas Hart, PhD, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Papworth Hospital, Cambridge
  - St James' University Hospital, Leeds
  - Guy's & St Thomas' NHS Foundation Trust, London
  - King's College Hospital, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Royal Free Hospital / University College London, London
  - John Radcliffe Hopsital, Oxford

REFERENCES:
- [Derived] Murphy PB, Brueggenjuergen B, Reinhold T, Gu Q, Fusfeld L, Criner G, Goss TF, Hart N. Cost-effectiveness of home non-invasive ventilation in patients with persistent hypercapnia after an acute exacerbation of COPD in the UK. Thorax. 2023 May;78(5):523-525. doi: 10.1136/thorax-2022-219653. Epub 2023 Feb 23. PMID 36823164
- [Derived] Murphy PB, Rehal S, Arbane G, Bourke S, Calverley PMA, Crook AM, Dowson L, Duffy N, Gibson GJ, Hughes PD, Hurst JR, Lewis KE, Mukherjee R, Nickol A, Oscroft N, Patout M, Pepperell J, Smith I, Stradling JR, Wedzicha JA, Polkey MI, Elliott MW, Hart N. Effect of Home Noninvasive Ventilation With Oxygen Therapy vs Oxygen Therapy Alone on Hospital Readmission or Death After an Acute COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2017 Jun 6;317(21):2177-2186. doi: 10.1001/jama.2017.4451. PMID 28528348